CLINICAL TRIAL: NCT00789490
Title: Relative Bioavailability of Iron and Folic Acid From a New Powdered Supplement Compared to a Traditional Tablet in Pregnant Women
Brief Title: Relative Bioavailability of Iron and Folic Acid in New Test Supplement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: The Hospital for Sick Children (Other); Heinz Endowments (Other)
Responsible Party: Dr Stanley Zlotkin M.D, PhD, FRCP (C), The Hospital For Sick Children
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Sickkids REB 1000007811
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Iron Deficiency; Folic Acid Deficiency
Keywords: pregnancy; relative bioavailability; iron; folic acid; ferric pyrophosphate; Study focus is to compare the relative bioavailability of SuppleFem Sprinkles to the current tradtional tablet Materna in pregnant women
MeSH Terms: conditions — Iron Deficiencies; Folic Acid Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Daminaide 995 - SuppleFem Sprinkles — The study agent SuppleFem will be a preblend manufactured by Acatris in Oakville Ontario and will be repackaged into 1 gram aliquots in white plastic Tamper Seal Vials.1 ram to be taken with test meal
Dietary Supplement: Materna — Materna is a pregnancy supplement available on the Canadian market and is manufactured by Wyeth. Dose is 1 tablet per day

SUMMARY:
Deficiencies of iron and folic acid during pregnancy can lead to adverse outcomes for the fetus, thus supplements are recommended. Adherence to current tablet-based supplements is documented to be poor. Recently a powdered form of micronutrients has been developed which may decrease side-effects and thus improve adherence. However, before testing the efficacy of the supplement as an alternate choice for supplementation during pregnancy, the bioavailability of the iron needs to be determined. The objective of this study is to measure the relative bioavailability of iron and folic acid from a powdered supplement that can be sprinkled on semi-solid foods or beverages versus a traditional tablet supplement in pregnant women.

DETAILED DESCRIPTION:
Background:

The proposal addresses the issue of the bioavailability of the supplement SuppleFem as compared to the current standard supplement Materna during pregnancy in Canadian women. In recognition of the difficulties Canadian women face in order to meet their iron (27 mg/day) and folic acid (600 µg/day) requirements from dietary sources alone during pregnancy, Health Canada currently recommends that an iron/folic acid supplement be taken by all women during pregnancy. However, because of issues related to adherence, many pregnant women do not fulfill the Health Canada recommendation. Adherence is largely influenced by the gastrointestinal side-effects associated with the use of iron tablets or pills, as well as the nausea and vomiting common during the first trimester. It is estimated that approximately10% of women discontinue the use of iron because of adverse effects while others use less than a daily dose. Women suffering from indigestion and heart-burn (gastro-esophageal acid reflux) associated with the use of iron supplements commonly discontinue their use and many find it difficult to swallow pills when nauseated.

The bioavailabilities of iron and folic acid in supplements may be an area of concern, primarily due to the higher requirements during pregnancy. Materna® contains a large quantity of calcium (250 mg), whereas Sprinkles contains none. A study by Hallberg, et al. (1991) showed that adding as little as 165 mg of calcium to a meal reduced the absorption of iron by 50-60% in wheat rolls. In addition, a study by Koren, et al. (2004) showed that after adjusting for dose, the iron absorbed from one maternal iron supplement containing calcium was statistically less as compared to one without calcium. A study by Rossander-Hultén et al (1991, as cited by Sandröm, 2001) found that zinc has the potential to inhibit iron absorption in supplements but not when zinc is added to food . The iron supplement contains 25mg of zinc whereas SuppleFem contains only 5.5mg. There are no reported interactions between folate and other nutrients. However, there is evidence that folate bioavailability may be influenced by the amount ingested. While pregnancy does increase the demand for folate, the amount in SuppleFem is compliant with the current DRI guidelines at 600µg, whereas the iron supplement contains 1000 µg. Currently, there is not enough research to indicate whether unmetabolized folic acid poses any health risks .

Rationale:

A new natural health product, "SuppleFem Sprinkles", was designed to address the issues with adherence. Sprinkles are single-dose sachets (like small packets of sugar) containing micronutrients in a powder form (iron as ferric pyrophosphate, folic acid and other micronutrients), which are easily sprinkled onto any foods or liquids prepared in the household. Any semi-solid food or liquid can be fortified by their addition. Sprinkles are meant to be added once daily to any semi-solid foods eaten in the home (eg: pureed fruits, orange juice or oatmeal), or mixed into a liquid. The efficacy of Sprinkles to prevent anemia in pregnant women has not previously been demonstrated, however, in the past five years, seven community-based trials in four different countries have examined the efficacy of Sprinkles in both infants and young children in developing countries xii, xiv, , , , , Before adherence can be measured as a primary outcome, however, it must be shown that there is no significant difference in the bioavailability of the ferric pyrophosphate in the SuppleFem® compared to the iron in the leading iron supplement thus showing that SuppleFem is as efficacious as standard treatments. If the new delivery system proves to be non-inferior to the leading iron tablets, then adherence to this new natural health product can be examined at a later date.

Trial Objectives:

Primary objective- The primary objective of this study is to determine whether or not the powdered formulation of micronized ferric pyrophosphate in SuppleFem® (to be mixed with liquids or food) is as bioavailable as the iron in the standard recommended pregnancy supplement.

Secondary Objective- The secondary objective of this study is to compare the relative bioavailability (ratio of AUCs for serum folate over an 8 hour period) of folic acid following a single dose of Materna® or Sprinkles.

Study Design & Duration:

The crossover design of the study will allow each subject to act as their own control. Since the interventions will be given in therapeutic dosage rather than a larger pharmaceutical dose it is anticipated that there should be no carryover effect to the next intervention. The washout periods between treatments will be one week each. It is anticipated that the study will begin September 1, 2005 and would last for a period of 6 to 9 weeks. Duration of study for each subject will be 3 weeks. Patients will be enrolled in the trial upon their answering of a posted advertisement. During the initial encounter, the prospective subjects will be informed as to the purpose of the trial, how the trial will be conducted, what their time commitment will be and any possible potential for harm This information will be explained by the study coordinator and informed consent will be obtained if the patient is agreeable. Subjects will fill out a baseline questionnaire detailing their supplement use as well as other demographic information before commencing the study. Prior supplement use should not impact on the relative bioavailability of either supplement since the crossover design will ensure prior use will impact on both treatments equally. Visit number one will determine diurnal variation values for the serum iron as well as establish iron status. Individuals in each of the groups will then be randomly allocated to either SuppleFem® or Materna® by selecting coloured poker chips from a bag to assign equal probability for each subject to fall into either of the two treatments. Two colors will be chosen to represent the two interventions. The chips will be placed in an opaque bag by the study coordinator and subjects will be asked at the commencement of the second visit (first intervention) to withdraw a chip from the bag as part of the randomization process. The colour will identify which intervention group the subject will be placed in. For visit number three, subjects will receive the opposite treatment from the one they took in visit two. Subject blinding is not possible due to the physical forms of the interventions; Materna is a large pill whereas Sprinkles are a granular powder. This study will be highly controlled and subjects will be closely observed while ingesting the supplements to ensure that the entire precisely measured amount is consumed. Further, serum measurements are objective in nature and cannot be influenced by the subject.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women between 18 and 45 years of age in the second or third trimester of pregnancy (24-32 weeks of gestational age).
* Normal Hb (Hb≥110g/L and Hb≤144g/L)

Exclusion Criteria:

Chronic illness (clinically significant neurological, endocrine, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic diseases)

* A history or presence of hemosiderosis, hemochromatosis, peptic ulcer, regional enteritis, ulcerative colitis
* A history of or current use of IV iron therapy or erythropoietin therapy
* A history or presence of any clinically significant gastrointestinal pathology (eg. chronic diarrhea, inflammatory bowel disease, partial gastrectomy), unresolved gastrointestinal symptoms (eg. diarrhea or vomiting), steatorrhea, or other conditions known to interfere with the absorption, distribution, metabolism or excretion of iron or folic acid
* Abnormal hemoglobin electrophoresis ie. sickle cell anemia, thalassemia, etc.
* Current acute illness and/or taking antibiotics
* Known or suspected allergies to Materna®, or any ingredient present in Materna or SuppleFem Sprinkles or any of the foods to be consumed during the trial.
* Mildly to severely anemic women (Hb<110 g/L) or elevated hemoglobin (above 144g/L)
* Complications in pregnancy (including pregnancy induced hypertension, preeclampsia, a history of severe antepartum hemorrhage)
* Blood transfusion within last 3 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a comparison of area under the curve (AUC) for change in serum iron for each intervention adjusted for diurnal variation. The use of AUC will provide a single outcome for each participant. | 3 weeks

SECONDARY OUTCOMES:
The secondary outcome is a comparison of area under the curve (AUC) for change in serum folate for each intervention | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital For Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hartman-Craven B, Christofides A, O'Connor DL, Zlotkin S. Relative bioavailability of iron and folic acid from a new powdered supplement compared to a traditional tablet in pregnant women. BMC Pregnancy Childbirth. 2009 Jul 27;9:33. doi: 10.1186/1471-2393-9-33. PMID 19635145